CLINICAL TRIAL: NCT03583814
Title: Rhode Island Asthma Integrated Response Program
Acronym: RI-AIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: State of Rhode Island Department of Health (Unknown); Providence Public School District (Unknown); Pawtucket School Department (Unknown); Central Falls School District (Unknown); Cranston Public Schools (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01HL138677 (NIH)
Record Dates: First submitted 2018-05-01; First posted 2018-07-11 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-04

CONDITIONS: Asthma in Children

STUDY DESIGN:
Intervention Model Description: The overall study utilizes a stepped wedge trial design with cluster randomization at the community level. All communities will have a baseline "control" period, active trial phase, and post-active trial phase follow-up period. During the active trial phase of this project, the strategy used to assign interventions to participants follows a Parallel Assignment study intervention model. During the active trial phase, individuals within that community will be assigned to an asthma intervention (1. CASE or 2. CASE and HARP) based on the child's level of asthma control. The SWT also allows us to compare community-level outcomes for participants who are not in the Active Trial (Intervention) period at that time and who are receiving standard care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CASE Program only (Active Comparator): During the Active Trial Phase, families of children with asthma status defined as "not well controlled" will complete the CASE program. Outcomes for participants assigned to the CASE program will be compared in a pre-post within subject comparison. Regardless of intervention arm assignment, children are expected show improvement in asthma outcomes. The stepped wedge trial design of the overall study allows for comparison of outcomes of communities in the pre-active trial baseline "control" period, active trial phase, and post-active trial phase follow-up period.
  Interventions: Behavioral: CASE Program
- CASE and HARP Programs (Active Comparator): During the Active Trial Phase, families of children with asthma status that is defined as "poorly controlled" will complete the CASE and HARP programs. Outcomes for participants assigned to this arm (CASE and HARP) will be compared in a pre-post within subject comparison. Regardless of intervention arm assignment, children are expected show improvement in asthma outcomes. The stepped wedge trial design of the overall study allows for comparison of outcomes of communities in the pre-active trial baseline "control" period, active trial phase, and post-active trial phase follow-up period.
  Interventions: Behavioral: CASE Program; Behavioral: HARP Program
- Standard Care (No Intervention): Cluster-based randomization in the Stepped Wedge Trial allows for comparison of Community Based Outcomes for clusters (communities defined by school catchment areas) who are not yet in the active trial phase and are receiving Standard of Care at that time.

INTERVENTIONS:
Behavioral: CASE Program — Controlling Asthma in Schools Effectively (CASE) provides school-based education and environmental assessments. This program takes place over the course of about 4 weeks and involves in-school or remote asthma education for school aged children, after-school or remote education sessions for their parents, asthma care training for school staff, and an evaluation of asthma triggers in the school.
  Arms: CASE Program only; CASE and HARP Programs
Behavioral: HARP Program — Home Asthma Response Program (HARP) is a home-visiting program consisting of 3 home visits or remote sessions (over about 6 weeks). HARP provides individualized asthma education, home-based environmental assessment, and strategies and supplies for controlling environmental asthma triggers.
  Arms: CASE and HARP Programs

SUMMARY:
The study's purpose is to evaluate the RI-Asthma Integrated Response (RI-AIR) Asthma Care Implementation Program (ACIP). RI-AIR ACIP uses an electronic information system to screen children with asthma and identify what specific services each child needs based on the child's asthma symptom and health care status. Our main goal is to see if children experience better asthma outcomes as a result of participation in the program. We will provide our intervention to 434 urban, ethnically diverse children, between 2-12 years old with asthma, and their families and evaluate whether participating in the program improves children's asthma outcomes. The second goal is to evaluate how well the program is set up and how we can make improvements to better serve families of children with asthma. The third goal is to gather information and advice from community experts so that we can make the program sustainable.

Families that take part in RI-AIR ACIP will participate in the program over the course of a year, including participating in the intervention, and brief follow up visits at 3, 6, 9 and 12 months after completing the intervention. All families will complete the CASE program, which takes place over the course of about 4 weeks and involves in-school or remote school-based asthma education for school aged children, after-school or remote education sessions for their parents, asthma care training for school staff, and an evaluation of asthma triggers in the school. Families of children who have more frequent asthma symptoms and emergency healthcare visits will also compete the HARP program, a home-based program consisting of 3 home sessions (over about 6 weeks) that include individualized asthma education and strategies and supplies for controlling environmental asthma triggers. Both CASE and HARP programs are carried out by certified asthma educators and community health workers.

Each child's healthcare provider (HCP) and school nurse teacher (SNT) will receive a standardized, secure email indicating the child is participating in RI-AIR. This email will include a summary of the child's baseline assessment of asthma control and prior health care use, and a description of the program. At the conclusion of the child's participation, the HCP and SNT will receive a summary by secure email summarizing the child's asthma control at the end of the intervention, services delivered, and referrals made, and for HARP participants, triggers observed in the home and supplies and referrals provided.

DETAILED DESCRIPTION:
The RI-AIR ACIP is community-based; it addresses community needs and gaps in care by: 1) enhancing asthma outcomes with services tailored to the child's level of asthma risk, 2) decreasing family burden by delivering services in homes and the local community, 3) enhancing communication between school, HCPs, and family, and 4) utilizing the RI-AIR Information Data System (IDS) to integrate data sources and generate a tailored referral. This study uses a randomized, stepped wedge trial (SWT) design to evaluate the effectiveness of the RI-AIR ACIP at both the individual and community levels. In an SWT, groups of individuals receive the intervention at different time points, the order in which they receive the treatment is randomized, and data are collected from groups over time.

In this study, groups will be randomized at the community level. Selected high risk communities are geographic school catchment areas with the highest asthma utilization rates. High-risk areas will be randomly allocated to the "Step," or year of active trial using a random numbers table. Thus, the year each catchment area receives intervention (i.e., participates in the active trial phase) will be randomized, and all families in this SWT will participate in both control (standard care) and intervention (active trial). This SWT design allows us to evaluate both individual-level outcomes as well as community-specific outcomes. During the active trial phase, families of children with asthma within the randomly selected communities will receive an asthma intervention. Families of children with asthma will be assigned to an intervention based on the child's level of asthma control. Individual-level data will be assessed over the course of the year of the active trial phase, while community-level data will be assessed annually over the study period.

ELIGIBILITY:
Inclusion Criteria:

* Child age between 2 to 12 years
* Child lives in the identified catchment area
* Child meets screening criteria for current asthma
* Child's asthma status is not well-controlled or poorly controlled
* Caregiver must speak English or Spanish.

Exclusion Criteria:

* Children with complex medical conditions (i.e., requiring on-site medical supervision of CHW)

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 432 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Asthma Control (Individual-Level) | During Active Trial Period at Baseline, End of Treatment (EOT; which will occur between 1 to 2 months after baseline, depending on intervention assignment), 3 month follow-up after EOT, 6 month follow-up, 9 month follow-up, 12 month follow-up
  Assessed by the Test for Respiratory and Asthma Control in Kids (TRACK) for 2-4 yr olds.
Change in Asthma Control (Individual Level) | During Active Trial Period at Baseline, End of Treatment (EOT; which will occur between 1 to 2 months after baseline, depending on intervention assignment), 3 month follow-up after EOT, 6 month follow-up, 9 month follow-up, 12 month follow-up
  Assessed by the Childhood Asthma Control Test (cACT) for 5-12 yr olds.

SECONDARY OUTCOMES:
Change in Asthma Symptom Free Days (Individual-Level) | During Active Trial Period at Baseline, End of Treatment (EOT; which will occur between 1 to 2 months after baseline, depending on intervention assignment), 3 month follow-up after EOT, 6 month follow-up, 9 month follow-up, 12 month follow-up
  Assessed by parent report using the standard questionnaire item, Symptom Free Days (SFDs) within previous 30-day period (Kirshnan et al., 2012). Parents are asked on how many days of the past 30 their child experienced asthma symptoms. This item is reverse-scored. Responses range from 0 to 30, with higher numbers indicating better functioning.
Change in caregivers' asthma self-efficacy, or their beliefs about how effectively they can manage their child's asthma (Individual-Level) | During Active Trial Period at Baseline, End of Treatment (EOT; which will occur between 1 to 2 months after baseline, depending on intervention assignment), 12 month followup after EOT
  Caregiver report of Asthma Management Efficacy. The Parent Asthma Self Efficacy Scale (Bursch et al., 1999) measures parents' self-efficacy with regard to managing their children's asthma. This questionnaire yields a total self-efficacy score, as well as scores for 2 subscales: Attack Prevention and Attack Management. Scores are derived by computing means of the items comprising that scale. Scores range from 1 to 5 with higher scores indicating higher parental self efficacy.
Change in Quality of Life related to Asthma as defined by the physical and emotional impact related to managing a child's asthma on the parent or caregiver (Individual-Level) | During Active Trial Period at Baseline, End of Treatment (EOT; which will occur between 1 to 2 months after baseline, depending on intervention assignment), 3 month followup after EOT, 6 month followup, 9 month followup, 12 month followup
  The Pediatric Asthma Caregiver's Quality of Life (QOL) Questionnaire (Juniper et al., 1996) assesses parent/caregiver's quality of life related to their children's asthma. This questionnaire yields a total score (overall QOL) as well as subscales related to parent's emotional functioning and activity functioning related to their child's asthma. The total score and subscales are each derived by computing a mean of the items comprising that scale. Scores range from 1 to 7 with higher scores indicating higher QOL.
Changes in health care utilization rates (Individual-level) | During Active Trial Period at Baseline and 12 month follow-up
  Assessed through electronic health record review of emergency department and inpatient visits
Changes in school absences (individual level) | During Active Trial Period at Baseline and 12 month follow-up
  Parent report of child's school absences
Changes in Asthma Health Care Utilization (Community-Level) | 12 months pre- and post-intervention year
  Community-based assessment of health care utilization using rates of emergency department visits and hospitalization for asthma from hospital data
Changes in number of School Absences (Community-Level) | 12 months pre- and post-intervention year
  Information from schools regarding children's school attendance across the academic year.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth L McQuaid, PhD, Principal Investigator — Rhode Island Hospital; Daphne Koinis Mitchell, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Following the NIH data sharing policy (2015), within one year of completion of the studies and dissemination of primary study results, public-use analysis datasets will be made available to the public, along with the final version of the study protocol, data dictionaries, and brief instructions. De-identification for the analysis datasets will follow published guidelines for "limited access data sets" funded by NHLBI (Geller et al., 2004).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available within one year of completion of the studies and dissemination of primary study results, and will be available for 10 years following the completion of the study.
Access Criteria: Once they become available, researchers requesting the data would follow the published RI-AIR ACIP procedures. We will make the data available to potential users only under a NIH-approved data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant in any way; (2) a commitment to securing the data using appropriate information security that is compliant with the most recent federal guidelines that are outlined by our information security protocol; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Cushman GK, Koinis-Mitchell D, Alsina M, Barker D, Drew L, DeCesare C, Yeo AJ, Durkin K, Elwy AR, Jandasek B, Pearlman DN, Vivier P, McQuaid EL. Design of a community-based, Hybrid Type II effectiveness-implementation asthma intervention study: The Rhode Island Asthma Integrated Response (RI-AIR) program. Contemp Clin Trials. 2023 Jun;129:107204. doi: 10.1016/j.cct.2023.107204. Epub 2023 Apr 23. PMID 37088129
- [Derived] McQuaid EL, Barker D, Chen ES, Coutinho MT, Cushman GK, Drew L, Elwy AR, Esteban CA, Jandasek BN, Kopel SJ, Pearlman D, Seifer R, Vivier P, Koinis-Mitchell D. Addressing Pediatric Asthma Disparities through RI-AIR's Community Approach: A Randomized Trial. Ann Am Thorac Soc. 2025 Nov;22(11):1709-1719. doi: 10.1513/AnnalsATS.202501-016OC. PMID 40569168